CLINICAL TRIAL: NCT00903136
Title: Screening for Barrett's Esophagus With an Ultrathin Scanning Fiber Endoscope
Brief Title: Tethered Capsule Endoscope in Screening Participants for Barrett Esophagus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Jason A. Dominitz, Veterans Affairs Medical Center - Seattle
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Screening
Other Study IDs: CDR0000641937; VAMC-WA-33141
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2010-02

CONDITIONS: Esophageal Cancer; Precancerous Condition
Keywords: Barrett esophagus; esophageal cancer; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Precancerous Conditions; Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Endoscopy, Digestive System; Endoscopy

INTERVENTIONS:
Other: questionnaire administration
Procedure: comparison of screening methods
Procedure: diagnostic endoscopic procedure
Procedure: esophagogastroduodenoscopy
Procedure: tethered capsule endoscopy

SUMMARY:
RATIONALE: A tethered capsule endoscope may be as effective as standard sedated endoscopy of the esophagus, stomach, and duodenum in screening for Barrett esophagus.

PURPOSE: This phase I/II trial is studying how well a tethered capsule endoscope works in screening participants for Barrett esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the clinical feasibility of obtaining endoscopic esophageal images using a tethered capsule endoscope (TCE). (Phase I)
* To determine the optimal weight and possibly shape for rapid patient ingestion and extraction of the TCE. (Phase I)
* To determine the optimal tether design (e.g., rigidity, distance markings, and other material properties). (Phase I)
* To determine the optimal protocol for patient ingestion and extraction of the TCE. (Phase I)
* To compare the TCE to standard sedated esophagogastroduodenoscopy for identifying suspected Barrett esophagus. (Phase II)

OUTLINE:

* Phase I: Participants swallow the tethered capsule endoscope (TCE) so that the distal end of the TCE enters the stomach. The TCE is then slowly withdrawn by the physician in order to visualize the gastroesophageal junction and the esophagus in a retrograde fashion until the upper esophageal sphincter is reached. The image acquisition process is repeated and the participant may be asked to swallow the TCE in up to 7 different positions with 2 swallows per position (no more than 20 swallows total).
* Phase II: Participants undergo TCE as in phase I, followed by standard sedated esophagogastroduodenoscopy (EGD) by a second physician.

Images obtained via TCE and EGD are reviewed by a third physician blinded to the results of each exam.

In both phases, participants and physicians complete a questionnaire after the TCE procedure to determine the ease of the procedure. Participants are also asked for specific suggestions to improve the TCE experience. Participants enrolled in phase II also complete a questionnaire 1 week after EGD to compare the TCE procedure with the EGD.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Healthy participant (phase I)
  * Scheduled to undergo esophagogastroduodenoscopy at the VA Puget Sound Health Care System for the evaluation of reflux symptoms (including screening for Barrett esophagus [BE]) or for follow-up of known BE (phase II)
* No current diagnosis of cancer

PATIENT CHARACTERISTICS:

* Not pregnant
* Able to fast for ≥ 6 hours prior to scheduled appointment
* No symptoms of dysphagia
* No history of a swallowing disorder (e.g., scleroderma, achalasia, esophageal stricture, or esophageal diverticulum)
* No history of a known or suspected gastrointestinal (GI) obstruction
* No other major medical illnesses (e.g., unstable cardiovascular disease, end-stage liver or kidney disease, or suspected active GI bleeding)
* No major physical disability that would prevent the participant from transferring from a chair to a bed and sitting up
* Not planning to undergo an MRI within 2 weeks after the study procedure

PRIOR CONCURRENT THERAPY:

* No prior surgery on the oropharynx, neck, esophagus, or stomach
* No concurrent anticoagulant medications or clopidogrel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Time required for swallowing the tethered capsule endoscope (TCE) to the stomach (Phase I)
Time required to image the squamo-columnar junction (Phase I)
Number of repeated swallows to achieve esophageal imaging (Phase I)
Amount of simethicone needed to reduce bubbles (Phase I)
Need for effervescent granules or other approaches to distend the esophagus (Phase I)
Time required for the entire TCE procedure (Phase I)
Quality of images (clarity, color, field of view, and resolution) obtained in the entire TCE procedure (Phase I)
Overall comfort during ingestion, pullback, and withdrawal of the TCE (Phase I)
Sensitivity, specificity, and accuracy of the TCE for identifying suspected Barrett esophagus (Phase II)
Agreement between the findings on the live TCE exam with the recorded TCE exam (Phase II)
Time to perform the TCE exam (Phase II)
Test characteristics of the first half vs the last half of the TCE exams performed by each of the 2 endoscopists (Phase II)
Comparison of participants' satisfaction with the TCE vs esophagogastroduodenoscopy (Phase II)

SECONDARY OUTCOMES:
Ability of the TCE to identify the presence or absence of other esophageal lesions (e.g., inflammation, diverticula, or varices) (Phase II)
Results of the histologic analysis of any biopsy specimens (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Jason A. Dominitz, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- Veterans Affairs Medical Center - Seattle, Seattle, Washington, United States